CLINICAL TRIAL: NCT00525044
Title: Double-blind, Randomized, Placebo-controlled Trial to Investigate the Efficacy and Tolerance of Ambroxol Lozenges 20 mg in the Treatment of Sore Throat in Patients With Acute Viral Pharyngitis
Brief Title: Double-blind Trial to Investigate Efficacy and Tolerance of Ambroxol Lozenges 20 mg in Sore Throat
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 18.490
Record Dates: First submitted 2007-09-03; First posted 2007-09-05 (Estimated); Results first posted 2019-07-11 (Actual); Last update posted 2019-07-11 (Actual); Status verified 2019-04

CONDITIONS: Pharyngitis
MeSH Terms: conditions — Pharyngitis | interventions — Ambroxol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Control (Placebo Comparator)
  Interventions: Drug: Placebo
- Ambroxol (Experimental)
  Interventions: Drug: Ambroxol

INTERVENTIONS:
Drug: Ambroxol
  Arms: Ambroxol
Drug: Placebo
  Arms: Control

SUMMARY:
The aim of this trial is to investigate the efficacy and tolerance of Ambroxol lozenges 20 mg in the treatment of sore throat in patients with acute viral pharyngitis.

DETAILED DESCRIPTION:
Male and female ambulant patients complaining of a sore throat caused by acute viral pharyngitis. Every patient may be included in the trial only once. A total of 250 male and female ambulant patients between the ages of 18 and 65 years will be enrolled. Approximately 8 centers will be recruited each enrolling approximately 30-32 patients.

Study Hypothesis:

The two-sided test hypothesis, that the results of the active treatment group with 20 mg Ambroxol and the placebo group do not differ with regard to the primary endpoint (null hypothesis (H0) will be tested against the alternative (H1) that they are not equal.

Comparison(s):

PRIMARY ENDPOINT:

Indication of pain on the VRS (PI)-verbal rating scale (pain intensity)-in the first 3 hours (the patient rates his/her pain on a six-point verbal rating scale).

SECONDARY ENDPOINT (S):

1. Patient's assessment of effectiveness and tolerance. The patient assesses the effectiveness and the tolerance of the test medicine for treating his sore throat at the end of the first and second day of treatment, by means of a verbal rating scale.
2. Participating doctors assessment of tolerance.

ELIGIBILITY:
1. Patients having a sore throat with acute viral pharyngitis. 2. Female and male ambulant patients between the ages of 18 and 65. 3. The throat pain intensity is rated at least severe on the VRS (PI). 4. Written Informed Consent is given by the patient. 5. Compliance by the patient seems guaranteed.

1. Patients with symptoms of primarily bacterial pharyngitis or bacterial secondary infection (clinical findings; inter alia assessment of exudate).
2. First indication of symptoms of acute pharyngitis (e.g., sore throat) occurred more than 3 days ago already.
3. Counting of white blood cell in blood routine examination exceeds 10?109/L.
4. Patients who suffered from acute viral or bacterial pharyngitis in the past 4 weeks.
5. Broncho-motor disorders or concomitant diseases with relatively large quantities of secretion (danger of secretion blockage).
6. Known hypersensitivity to Ambroxol or to auxiliary substances contained in the tablet.
7. Previous and/or existing tumour condition.
8. Pregnancy and/or breast-feeding.
9. Alcohol, and/or drug abuse.
10. Simultaneous participation in another clinical trial.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2007-08-01 (Actual); Primary Completion 2008-01-01 (Actual); Study Completion 2008-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — Boehringer Ingelheim Shanghai
Locations (4):
- China (4):
  - Boehringer Ingelheim Investigational Site, Nanjing
  - Boehringer Ingelheim Investigational Site, Shanghai
  - ENT Subsidiary of Fudan University Hospital, Shanghai
  - Boehringer Ingelheim Investigational Site, Wuhan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Male or female outpatients, 18 to 65 years of age, suffering from acute viral pharyngitis and throat pain of at least severe intensity were to enter the trial.
Pre-assignment Details: Double-blind, randomized, placebo-controlled parallel design in comparison of two arms
Groups:
- Ambroxol Lozenges 20 mg: Patients were orally administered Ambroxol lozenges 20 milligram (mg) initially (first lozenges); up to 6 lozenges per day up to two days, maximal dose:120 mg per day
- Placebo: Patients were orally administered Placebo matching Ambroxol lozenges 20 mg initially (first lozenges); up to 6 lozenges per day up to two days.
Period: Overall Study
Arm/Group | Ambroxol Lozenges 20 mg | Placebo
Started | 124 | 125
Completed | 124 | 124
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): FAS, which included all patients
  * who were randomized,
  * who took at least the first lozenge,
  * who had Pain Intensity (PI) data of baseline.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ambroxol Lozenges 20 mg | Placebo | Total
Number analyzed (Participants) | 124 | 125 | 249
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.0 (12.2) | 38.4 (13.0) | 37.2 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 71 | 138
  Male | 57 | 54 | 111

OUTCOME MEASURES:

1. Primary Outcome: Sum of Pain Intensity Difference (SPIDnorm)-Time-weighted Average of the Pain Intensity Difference (PID) From Pre-dose Baseline Over the First 3 Hours After the First Lozenge Expressed as a Ratio of the Pre-dose Baseline
Description: The calculation will be based on the pain intensity (PI) assessment by the patient before and then at (pain intensity difference at 30 minutes (PID30)), (pain intensity difference at 60 minutes (PID60)), (pain intensity difference at 120 minutes (PID120)) and (pain intensity difference at 180 minutes (PID180)) after the 1st lozenge. Using the difference in PI from pre-dose baseline for each time point subsequent to dosing, the SPIDnorm will be calculated as SPIDnorm = (30*PID30 + 30*PID60 + 60*PID120 + 60*PID180)/(180*PI (baseline)) The patient rates the intensity of his sore throat pain on a 6-point Verbal Rating Scale (VRS) pain intensity (PI) before taking the first lozenge and 30, 60, 120 and 180 minutes thereafter, and enters his rating in his patient's diary . The rating scale is as follows: 0=no pain; 1=hardly any pain; 2=slight pain; 3=moderate pain; 4=severe pain; 5=very severe pain.
Time Frame: pre-dose baseline and 30, 60, 120, and 180 minutes
Population: Full Analysis Set (FAS): FAS, which included all patients
  * who were randomized,
  * who took at least the first lozenge,
  * who had PI data of baseline.
Measure: Least Squares Mean (Standard Error); unit: ratio
Groups:
- Ambroxol Lozenges 20 mg: Patients were orally administered Ambroxol lozenges 20 mg initially (first lozenges); up to 6 lozenges per day up to two days, maximal dose:120 mg per day
Arm/Group | Ambroxol Lozenges 20 mg | Placebo
Number analyzed (Participants) | 124 | 125
ratio | -0.40 (0.020) | -0.34 (0.020)
Statistical Analysis 1: Comparison: Ambroxol Lozenges 20 mg vs Placebo; Differences between the treatment groups with regard to the primary endpoint SPIDnorm was tested using an analysis of variance (ANOVA) including treatment and centre as fix effects. Treatment differences were estimated by reference to the adjusted least squares mean differences and the corresponding 95 % confidence intervals; Test type: Other; p = 0.0156, ANOVA; Mean Difference (Final Values) = -0.07, 95% CI 2-sided [-0.12 to -0.01], Standard Error of Mean 0.028 — Treatment differences (Ambroxol- Placebo)

2. Secondary Outcome: Pain Intensity (PI) as Rated on a 6-point VRS by the Patient at 0.5, 1, 2 and 3 Hours After the First Lozenge
Description: Pain intensity (PI) as rated on a 6-point Verbal Rating Scale (VRS) by the patient at 0.5, 1, 2 and 3 hours after the first lozenge.
  The patient rates the intensity of his sore throat condition on a 6-point rating scale [VRS(PI)-verbal rating scale (pain intensity)] before taking the first lozenge and 30, 60, 120 and 180 minutes thereafter, and enters his rating in his patient's diary . The rating scale is as follows: 0=no pain; 1=hardly any pain; 2=slight pain; 3=moderate pain; 4=severe pain; 5=very severe pain.
  Adjusted Mean (Standard Error) are presented for this outcome measure.
Time Frame: 0.5, 1, 2 and 3 hours
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Ambroxol Lozenges 20 mg | Placebo
Number analyzed (Participants) | 124 | 125
score on a scale
  30 minutes | 2.9 (0.08) | 3.1 (0.07)
  60 minutes | 2.6 (0.08) | 2.8 (0.08)
  120 minutes | 2.3 (0.10) | 2.7 (0.09)
  180 minutes | 2.2 (0.10) | 2.5 (0.10)
Statistical Analysis 1: Comparison: Ambroxol Lozenges 20 mg vs Placebo; Analysis at 30 min: analysis of covariance (ANCOVA) including treatment and centre as fix effects and baseline as covariable are presented. Treatment differences are estimated by reference to the adjusted least squares mean differences and the corresponding 95 % confidence intervals; Test type: Other; p = 0.1280, ANCOVA; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.4 to 0], Standard Error of Mean 0.10 — Treatment differences (Ambroxol- Placebo)
Statistical Analysis 2: Comparison: Ambroxol Lozenges 20 mg vs Placebo; Analysis at 60 min: analysis of covariance (ANCOVA) including treatment and centre as fix effects and baseline as covariable are presented. Treatment differences are estimated by reference to the adjusted least squares mean differences and the corresponding 95 % confidence intervals; Test type: Other; p = 0.0417, ANCOVA; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.4 to 0.0], Standard Error of Mean 0.11 — Treatment differences (Ambroxol- Placebo)
Statistical Analysis 3: Comparison: Ambroxol Lozenges 20 mg vs Placebo; Analysis at 120 min: analysis of covariance (ANCOVA) including treatment and centre as fix effects and baseline as covariable are presented. Treatment differences are estimated by reference to the adjusted least squares mean differences and the corresponding 95 % confidence intervals; Test type: Other; p = 0.0054, ANCOVA; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-0.6 to -0.1], Standard Error of Mean 0.13 — Treatment differences (Ambroxol- Placebo
Statistical Analysis 4: Comparison: Ambroxol Lozenges 20 mg vs Placebo; Analysis at 180 min: analysis of covariance (ANCOVA) including treatment and centre as fix effects and baseline as covariable are presented. Treatment differences are estimated by reference to the adjusted least squares mean differences and the corresponding 95 % confidence intervals; Test type: Other; p = 0.0201, ANCOVA; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-0.6 to 0.0], Standard Error of Mean 0.13 — Treatment differences (Ambroxol- Placebo

3. Secondary Outcome: Pain Intensity Difference From Pre-dose Baseline (PID) as Rated on a 6-point Verbal Rating Scale (VRS) by the Patient at 0.5, 1, 2 and 3 Hours After the First Lozenge
Description: Pain intensity difference from pre-dose baseline (PID) as rated on a 6-point Verbal Rating Scale (VRS) by the patient at 0.5, 1, 2 and 3 hours after the first lozenge.
  Adjusted Mean (Standard Error) are presented for this outcome measure.
Time Frame: pre-dose baseline and 0.5, 1, 2 and 3 hours
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Ambroxol Lozenges 20 mg | Placebo
Number analyzed (Participants) | 124 | 125
score on a scale
  30 minutes | -1.1 (0.08) | -1.0 (0.07)
  60 minutes | -1.4 (0.08) | -1.2 (0.08)
  120 minutes | -1.8 (0.10) | -1.4 (0.09)
  180 minutes | -1.9 (0.10) | -1.6 (0.10)
Statistical Analysis 1: Comparison: Ambroxol Lozenges 20 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.1280, ANCOVA; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.4 to 0.0], Standard Error of Mean 0.10 — Treatment differences (Ambroxol- Placebo)
Statistical Analysis 2: Comparison: Ambroxol Lozenges 20 mg vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Other; p = 0.0417, ANCOVA; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.4 to 0.0], Standard Error of Mean 0.11 — Treatment differences (Ambroxol- Placebo
Statistical Analysis 3: Comparison: Ambroxol Lozenges 20 mg vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Other; p = 0.0054, ANCOVA; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-0.6 to -0.1], Standard Error of Mean 0.13 — Treatment differences (Ambroxol- Placebo
Statistical Analysis 4: Comparison: Ambroxol Lozenges 20 mg vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Other; p = 0.0201, ANCOVA; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-0.6 to 0.0], Standard Error of Mean 0.13 — Treatment differences (Ambroxol- Placebo

4. Secondary Outcome: Assessment of Redness of the Pharyngeal Mucosa by the Investigator on a 5-point VRS at Pre-dose Baseline and at the End-of-study Evaluation
Description: Assessment of redness of the pharyngeal mucosa by the investigator on a 5-point VRS (normal, slightly red, clearly red, very red, severe inflammation) at pre-dose baseline and at the end-of-study evaluation.
Time Frame: Day 1 and Day 2
Population: SAFETY Set, which included all patients
  * who were randomized,
  * who took at least one dose of trial medication.
Measure: Number; unit: percentage of participants
Arm/Group | Ambroxol Lozenges 20 mg | Placebo
Number analyzed (Participants) | 124 | 125
percentage of participants
  Day 1_Normal | 0.0 | 0.8
  Day 1_Slightly red | 12.1 | 12.8
  Day 1_ Clearly red | 53.2 | 50.4
  Day 1_Very red | 29.8 | 32.0
  Day 1_Severe inflammation | 4.8 | 4.0
  Day 2_Normal: number analyzed (Participants) | 124 | 124
  Day 2_Normal | 12.1 | 10.5
  Day 2_Slightly red: number analyzed (Participants) | 124 | 124
  Day 2_Slightly red | 66.9 | 66.9
  Day 2_Clearly red: number analyzed (Participants) | 124 | 124
  Day 2_Clearly red | 18.5 | 21.8
  Day 2_Very red: number analyzed (Participants) | 124 | 124
  Day 2_Very red | 2.4 | 0.8
  Day 2_Severe inflammation: number analyzed (Participants) | 124 | 124
  Day 2_Severe inflammation | 0.0 | 0.0
Statistical Analysis 1: Comparison: Ambroxol Lozenges 20 mg vs Placebo; Analysis at day 1: P-value was calculated by the Cochran-Mantel-Haenszel test adjusting for center; Test type: Other; p = 0.9939, Mantel Haenszel
Statistical Analysis 2: Comparison: Ambroxol Lozenges 20 mg vs Placebo; Analysis at day 2: P-value was calculated by the Cochran-Mantel-Haenszel test adjusting for center; Test type: Other; p = 0.5552, Mantel Haenszel

5. Secondary Outcome: Assessment of Patients' Assessment of Effectiveness on a 5-point VRS at Pre-dose Baseline and at the End-of-study Evaluation
Description: Assessment of Patients' Assessment of Effectiveness on a 5-point VRS ("very good", "good", "neither good nor poor", "not very good", "not at all good") at pre-dose baseline and at the end-of-study evaluation
Time Frame: Day 1 and Day 2
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | Ambroxol Lozenges 20 mg | Placebo
Number analyzed (Participants) | 124 | 125
percentage of participants
  Day 1_Very good | 13.7 | 8.0
  Day 1_Good | 58.1 | 52.0
  Day 1_Neither good nor poor | 19.4 | 18.4
  Day 1_Not very good | 6.5 | 16.0
  Day 1_Not at all good | 2.4 | 5.6
  Day 2_Very good: number analyzed (Participants) | 111 | 113
  Day 2_Very good | 24.3 | 14.2
  Day 2_Good: number analyzed (Participants) | 111 | 113
  Day 2_Good | 56.8 | 52.2
  Day 2_Neither good nor poor: number analyzed (Participants) | 111 | 113
  Day 2_Neither good nor poor | 14.4 | 16.8
  Day 2_Not very good: number analyzed (Participants) | 111 | 113
  Day 2_Not very good | 3.6 | 13.3
  Day 2_Not at all good: number analyzed (Participants) | 111 | 113
  Day 2_Not at all good | 0.9 | 3.5
Statistical Analysis 1: Comparison: Ambroxol Lozenges 20 mg vs Placebo; Analysis at day 1: P-value was calculated by the Cochran-Mantel-Haenszel test adjusting for center; Test type: Other; p = 0.0343, Mantel Haenszel
Statistical Analysis 2: Comparison: Ambroxol Lozenges 20 mg vs Placebo; Analysis at day 2: P-value was calculated by the Cochran-Mantel-Haenszel test adjusting for center; Test type: Other; p = 0.0119, Mantel Haenszel

ADVERSE EVENTS:
Time Frame: From drug administration until end of the treatment, up to 2 days.
Arm/Group | Ambroxol Lozenges 20 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/124 | 0/125
Serious Adverse Events (participants affected / at risk) | 0/124 | 0/125
Other Adverse Events (participants affected / at risk) | 0/124 | 0/125

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No